CLINICAL TRIAL: NCT04673370
Title: A Pilot Study of Ba Duan Jin for Depression and Anxiety
Brief Title: Ba Duan Jin for Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Lu Ying, MM, Research Associate, Shanghai University of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZY(2018-2020)-CCCX-2007
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A total of 60 patients were divided into a treatment group and a control group, with 30 cases in each group. The control group received health education，and the treatment group was treated with Ba Duan Jin plus health education program.
Who Masked: Outcomes Assessor
Masking Description: The study was a single-blind controlled trial in which the outcome assessor was blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ba Duan Jin Group (Experimental): Ba Duan Jin plus health education. Participants take part in 16-week program. The health education is conducted as the Health Education Group. Besides, the participants attended two 90-minute sessions of group-based Ba Duan Jin training per week and practiced at least three 30-minute Ba Duan Jin sessions at home per day.
  Interventions: Behavioral: Ba Duan Jin
- Health Education Group (Active Comparator): Health education. Participants take part in 16-week program. The health education includes work, rest, diet and other basic programs according to the different conditions of participants.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Ba Duan Jin — Ba Duan Jin, a traditional Chinese health-preserving technique, combines techniques regulating body, breath and spirit. According to traditional Chinese theory, every movement of Ba Duan Jin has unique effect to different Zang-fu organs.
  Other Names: Eight-section Brocade
  Arms: Ba Duan Jin Group
Behavioral: Health education — Health education is provided by psychologist and TCM doctor, including work, rest, diet and other basic programs.
  Arms: Health Education Group

SUMMARY:
In recent years, the number of people with symptoms of depression or anxiety are on the rise. The aims of the present study is to examine the effects of Ba Duan Jin on reducing symptoms of depression or anxiety.

DETAILED DESCRIPTION:
There is growing interest in mind-body therapy that could potentially improve patients' psychological health.

Ba Duan Jin, a traditional Chinese health-preserving technique, combines techniques regulating body, breath and spirit. The effects of Ba Duan Jin on patients with symptoms of depression and anxiety are yet to be further investigated.

The present pilot clinical study aims to apply Ba Duan Jin to patients with symptoms of depression and anxiety, and to evaluate the psychological effects.

Participants allocated to the Health Education Group take part in the 16-week health education including work, rest, diet and other basic programs according to the different conditions of participants. Participants allocated to the Ba Duan Jin Group take part in the 16-week Ba Duan Jin plus health education program. The study plans to enroll 60 participants (30 for Ba Duan Jin plus health education program, and 30 for health education program), expecting that Ba Duan Jin has a better effect on improving psychological condition.

ELIGIBILITY:
Inclusion Criteria:

* Subject with depression or anxiety symptom diagnosed by ICD-10.
* Subject is male or female, age 18 to 75.
* Subject has a clear mind and the ability to read, to talk and to communicate.
* Subject agrees to participate in this study and sign to the informed consent

Exclusion Criteria:

* Subject has severe somatic disease.
* Subject has history of organic mental disorder, epilepsy, schizophrenia.
* Subject takes any medication of food having effect on gut microbiota within 1 month of screening.
* Subject has history of alcohol abuse.
* Subject is pregnant, lactating or breast-feeding women.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Depression Rating Scale | Change from Baseline HAMD-17 at 16 weeks
  The HAMD-17 is a clinician-rated assessment (structured interview) of patients' depressive symptoms. Questions focus on depressive symptoms during the past 7 days, and higher cumulative scores indicate more severe depression.
14-item Hamilton Anxiety Rating Scale | Change from Baseline HAMA-14 at 16 weeks
  The HAMA-14 is a clinician-rated assessment (structured interview) of patients' anxious symptoms. Questions focus on anxious symptoms during the past 7 days, and higher cumulative scores indicate more severe anxiety.

SECONDARY OUTCOMES:
Depression, Anxiety and Stress Scale-21 item | Baseline
  The DASS-21 is a self-rated assessment of patients' depressive, anxious and stress symptoms. Questions focus on depressive, anxious and stress symptoms during the past 7 days, and higher cumulative scores indicate more severe depression, anxiety and stress. Subscale scores are calculated as the sum of the responses to the seven items from each subscale multiplied by 2. The cutoffs for depression, anxiety, and stress are >9, >7, and >14, respectively.
Depression, Anxiety and Stress Scale-21 item | 8 weeks
  The DASS-21 is a self-rated assessment of patients' depressive, anxious and stress symptoms. Questions focus on depressive, anxious and stress symptoms during the past 7 days, and higher cumulative scores indicate more severe depression, anxiety and stress. Subscale scores are calculated as the sum of the responses to the seven items from each subscale multiplied by 2. The cutoffs for depression, anxiety, and stress are >9, >7, and >14, respectively.
Depression, Anxiety and Stress Scale-21 item | 16 weeks
  The DASS-21 is a self-rated assessment of patients' depressive, anxious and stress symptoms. Questions focus on depressive, anxious and stress symptoms during the past 7 days, and higher cumulative scores indicate more severe depression, anxiety and stress. Subscale scores are calculated as the sum of the responses to the seven items from each subscale multiplied by 2. The cutoffs for depression, anxiety, and stress are >9, >7, and >14, respectively.
Gut microbiota | Baseline
  Intestinal microbiome in stool will be measured by 16S sequencing.
Gut microbiota | 16 weeks
  Intestinal microbiome in stool will be measured by 16S sequencing.
Traditional Chinese medicine syndrome grade | Baseline
  Traditional Chinese medicine(TCM) syndrome will be evaluated by TCM syndrome questionnaire.
Traditional Chinese medicine syndrome grade | 16 weeks
  Traditional Chinese medicine(TCM) syndrome will be evaluated by TCM syndrome questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Qigong Research Institute, Shanghai, Shanghai Municipality, China